CLINICAL TRIAL: NCT04564417
Title: Phase I Dose Escalation and Dose Expansion, International, Multicenter Study of W0180 as Single Agent and in Combination With Pembrolizumab (Anti-PD-1) in Adult Participants With Locally Advanced or Metastatic Solid Tumors
Brief Title: First-In-Human (FIH) Study of W0180 as Single Agent and in Combination With Pembrolizumab in Adults With Locally Advanced or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: W00180IV101; 2019-002299-15 (EudraCT Number)
Record Dates: First submitted 2020-08-31; First posted 2020-09-25 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-07

CONDITIONS: Locally Advanced or Metastatic Solid Tumors
Keywords: advanced cancer; W0180
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Monotherapy dose escalation: W0180 (Experimental): Participants will receive W0180 in a 21-day cycle until the maximum tolerated dose (MTD)/ recommended dose for expansion (RDE) for the single-agent identified.
  Interventions: Biological: W0180
- Combination dose escalation: W0180+Pembrolizumab (Experimental): Participants will receive Pembrolizumab 200 mg flat dose as IV infusion every three weeks (Q3W) followed by W0180 in a 21-day Cycle until the MTD in combination is identified or an RDE in combination is established.
  Interventions: Biological: W0180; Drug: Pembrolizumab
- Dose expansion (Experimental): Participants will receive Pembrolizumab 200 mg flat dose as IV infusion Q3W followed by an RDE dose of W0180 in a 21-day cycle.
  Interventions: Biological: W0180; Drug: Pembrolizumab

INTERVENTIONS:
Biological: W0180 — Participants will receive W0180 in a 21-day cycle.
Drug: Pembrolizumab — Participants will receive Pembrolizumab 200 mg flat dose as IV infusion every three weeks (Q3W) in a 21-day cycle.
  Arms: Combination dose escalation: W0180+Pembrolizumab; Dose expansion

SUMMARY:
The purpose of this study will be to determine the Maximum Tolerated Dose (MTD) and describe dose-limiting toxicities (DLTs) of W0180 given as monotherapy and in combination with pembrolizumab (anti-PD-1).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of locally advanced or metastatic solid tumors, whose disease has progressed or for whom no further standard therapy is available or appropriate
* Evidence of measurable disease as determined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (or modified RECIST 1.1 for mesothelioma)
* Adequate blood counts at baseline
* Adequate liver function at screening and baseline
* Sexually active participants must use medically acceptable methods of contraception during the course of this study

Exclusion Criteria:

* Participants previously treated with an anti-V-domain Ig suppressor of T cell activation (VISTA) (small molecule or antibody) agent
* Participants with known central nervous system (CNS) metastases and/or carcinomatous meningitis
* History of severe hypersensitivity reactions to other monoclonal antibodies
* Positive for hepatitis B virus(HBV), hepatitis C virus (HCV) or HIV infection
* History of anti-cancer therapies within the last 4 weeks (or <=5 half-lives for targeted agents) prior to initiating study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Dose-limiting Toxicities (DLTs) During the DLT Period | From Cycle 1-Day 1 up to Cycle 2-Day 1 (each cycle of 21 days)
  The DLTs will be classified according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.

SECONDARY OUTCOMES:
Escalation Part: Recommended Dose for Expansion After Administration of W0180 in Monotherapy and in Combination With Pembrolizumab | From the first study treatment infusion in Cycle 1 (each cycle of 21 days) until the safety follow-up in Combination dose escalation cohort (30 days after last study infusion administration) (approximately 22 months)
  The RDE will be the dose of W0180 chosen for the dose-expansion part.
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs) | From the first study treatment infusion in Cycle 1 (each cycle of 21 days) until the safety follow-up in expansion part (approximately 44 months)
  Treatment-Emergent Adverse Events (TEAEs)/Treatment-Emergent Serious Adverse Events (TESAEs) are any new event that starts after the first administration of study treatment and less than or equal to (<=) 30 days after treatment discontinuation or that worsened during that study period.
Number of Participants With Treatment-Emergent Adverse Events by Severity | From the first study treatment infusion in Cycle 1 (each cycle of 21 days) until the safety follow-up in expansion part (approximately 44 months)
  The severity of the AEs are categorized into Grades 1 to 5: Grade 1: Mild- asymptomatic or mild symptoms, Grade 2: Moderate- minimal; local or noninvasive intervention indicated, Grade 3: Severe or medically significant but not immediately life-threatening, Grade 4: Life-threatening consequences, and Grade 5: Death related to AE. An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. TEAE is any new event that starts after the first administration of study treatment and <=30 days after treatment discontinuation or that worsened during that study period.
Number of Participants With Clinically Significant Laboratory Abnormalities Reported as Treatment-Emergent Adverse Events (TEAE) | From the first study treatment infusion in Cycle 1 (each cycle of 21 days) until the safety follow-up in expansion part (approximately 44 months)
  Number of participants with clinically significant abnormalities in laboratory parameters (hematology, blood chemistry, coagulation parameters, thyroid function, urinalysis, cytokines and tryptase) will be assessed after administration of W0180 in monotherapy and in combination with pembrolizumab for both escalation and expansion part of study.
Number of Participants With Dose Interruptions, Dose Reductions, or Discontinuation After Administration of W0180 in Monotherapy and in Combination With Pembrolizumab | From the first study treatment infusion in Cycle 1 (each cycle of 21 days) until the safety follow-up in expansion part (approximately 44 months)
  The number of participants reporting dose interruptions, dose reductions, and temporary or definitive discontinuation after administration of W0180 in monotherapy and in combination with pembrolizumab for both escalation and expansion part of study will be assessed.
Duration of Study Drug Exposure in Participants | From the first study treatment infusion in Cycle 1 (each cycle of 21 days) until the safety follow-up in expansion part (approximately 44 months)
  The duration of study treatment exposure will be summarized after the administration of W0180 in monotherapy and in combination with pembrolizumab for both escalation and expansion part of the study.
Actual and Relative Dose Intensity in Participants | From the first study treatment infusion in Cycle 1 (each cycle of 21 days) until the safety follow-up in expansion part (approximately 44 months)
  Participants with actual and relative dose intensity will be summarized and assessed after administration of W0180 in monotherapy and in combination with pembrolizumab.
Escalation Part: Objective Response Rate (ORR/iORR) | Every 6 weeks for 12 months then every 8 weeks, until disease progression (Approximately 22 months)
  The ORR/iORR will be assessed and reported per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 and per immune Response Evaluation Criteria in Solid Tumors (iRECIST).
Escalation Part: Disease Control Rate (DCR) Assessed by RECIST | Every 6 weeks for 12 months then every 8 weeks, until disease progression (Approximately 22 months)
  The DCR will be assessed per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Escalation Part: Immune Disease Control Rate (iDCR) Assessed by iRECIST | Every 6 weeks for 12 months then every 8 weeks, until disease progression (Approximately 22 months)
  The iDCR will be assessed and reported per immune Response Evaluation Criteria in Solid Tumors (iRECIST).
Observed Maximum Plasma Concentration (Cmax) | From Cycle 1 Day 1 Predose to Cycle 8 Day 1: Predose (each cycle of 21 days)
  Cmax will be assessed after administration of W0180 in monotherapy and in combination with pembrolizumab.
Experimental Half-life (T1/2) | From Cycle 1 Day 1 Predose to Cycle 8 Day 1: Predose (each cycle of 21 days)
  T1/2 will be assessed after administration of W0180 in monotherapy and in combination with pembrolizumab.
Area Under the Plasma Concentration-time Curve From Zero to the Last Quantifiable Point (AUC0-t) | From Cycle 1 Day 1 Predose to Cycle 8 Day 1: Predose (each cycle of 21 days)
  AUC0-t will be assessed after administration of W0180 in monotherapy and in combination with pembrolizumab.
Total Clearance | From Cycle 1 Day 1 Predose to Cycle 8 Day 1: Predose (each cycle of 21 days)
  Total Clearance will be Calculated as the Ratio of the Dose and the total area under the plasma concentration-time curve (AUCinf). CLtot will be assessed after administration of W0180 in monotherapy and in combination with pembrolizumab.
Number of Participants With Anti-W0180 Antibodies Post Administration of W0180 as Monotherapy and in Combination With Pembrolizumab | From the first study treatment infusion in Cycle 1 (each cycle of 21 days) until the safety follow-up in expansion part (approximately 44 months)
Expansion Part: Objective Response Rate (ORR/iORR): Confirmed and Unconfirmed | Every 6 weeks for 12 months then every 8 weeks, until disease progression (Approximately 44 months)
  ORR/iORR will be assessed and reported per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 and per immune Response Evaluation Criteria in Solid Tumors (iRECIST).
Expansion Part: Duration of response (DOR/iDOR) | Every 6 weeks for 12 months then every 8 weeks, until disease progression (Approximately 44 months)
  The DOR/iDOR will be assessed and reported per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 and per immune Response Evaluation Criteria in Solid Tumors (iRECIST).
Expansion Part: Time to treatment response (TTR) | Every 6 weeks for 12 months then every 8 weeks, until disease progression (Approximately 44 months)
  The TTR will be assessed and reported per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 and per immune Response Evaluation Criteria in Solid Tumors (iRECIST).
Expansion Part: Progression Free Survival (PFS) Assessed per RECIST v1.1 | Every 6 weeks for 12 months then every 8 weeks, until disease progression (Approximately 44 months)
  The progression free survival will be assessed and reported per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Expansion Part: Progression-Free Survival (iPFS) Assessed per iRECIST | Every 6 weeks for 12 months then every 8 weeks, until disease progression (Approximately 44 months)
  The iPFS will be assessed and reported per immune Response Evaluation Criteria in Solid Tumors (iRECIST).
Expansion Part: Disease Control Rate (DCR) Assessed per RECIST v1.1 | Every 6 weeks for 12 months then every 8 weeks, until disease progression (Approximately 44 months)
  The DCR will be assessed and reported per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Expansion Part: Disease Control Rate (iDCR) Assessed per iRECIST | Every 6 weeks for 12 months then every 8 weeks, until disease progression (Approximately 44 months)
  The iDCR will be assessed and reported per immune Response Evaluation Criteria in Solid Tumors (iRECIST).
Expansion Part: Overall survival (OS) | Every 6 weeks for 12 months then every 8 weeks, until disease progression (Approximately 44 months)
  OS is defined as time duration which was measured from the date of first dose to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Locations (5):
- France (3):
  - Centre Leon Berard, department Medical Oncology, Lyon, Cedex
  - IUCT, Toulouse, Toulouse
  - IGR, Villejuif, Villejuif
- Spain (2):
  - CUN, Madrid, Madrid
  - CUN, Pamplona, Pamplona

IPD SHARING:
Plan to Share IPD: No